CLINICAL TRIAL: NCT06879639
Title: The Effect of 10 Weeks of Physical Exercise on Glycated Hemoglobin and Blood Pressure in Elderly People With Multimorbidity Conditions: a Controlled and Randomized Study
Brief Title: Exercise Impact in Elderly With Multimorbidity: HbA1c and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEFADE 27_2024
Record Dates: First submitted 2025-02-11; First posted 2025-03-17 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-01

CONDITIONS: Hypertension; Diabetes; Osteoarthritis; Depression Disorders; Multimorbidity; Respiratory Disorders; Sarcopenia in Elderly; Dyslipidemia; High Blood Cholesterol; Obese Patients
Keywords: Multimorbidity; Diabetes; High blood pressure; Older people; Combined exercise; Aquatic exercise
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Osteoarthritis; Respiration Disorders; Dyslipidemias | interventions — Exercise; Control Groups; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Combined physical exercise in land (Experimental): Combined physical exercise performed in gym 3 times per week
  Interventions: Other: Exercise
- Combined physical exercise in water (Experimental): Combined physical exercise performed in water 3 times per week.
  Interventions: Other: Exercise
- Control Group (Experimental): The control group will not performed physical exercise for ten weeks.
  Interventions: Other: Control

INTERVENTIONS:
Other: Exercise — The workout routine for the Land Exercise (LE) group will be segmented as follows: A cardio segment (15-20 minutes) involving treadmill walking/running or cycling on the stationary bike; A strength training segment (35 minutes) comprising bench press, seated row, leg extension, squats, pull down, peck-deck, hamstring curls, curl-ups, and back extensions; and a cool-down phase (5-10 minutes) featuring stretching exercises.
  Other Names: Physical exercise; Combined exercise
  Arms: Combined physical exercise in land
Other: Control — The control group will not receive any formal indication or support to perform structured exercise training but will be allowed to engage in physical activity ad libitum.
  Other Names: Control group; No intervention group
  Arms: Control Group
Other: Exercise — The activities for the Water Exercise (WE) group will be divided into segments: An aerobic portion (15-20 minutes) involving water walking and jogging combined with arm movements; A resistance portion (35 minutes) including chest/upper back guidance, chest back press, behind-the-back press, pivoted shoulder press (upper body), and calf lifts, supported squats, outer/inner thigh scissors, and forward and back leg glide (lower body), and finally, a cool-down period (5-10 minutes) comprising stretching exercises.
  Other Names: Combined exercise in water
  Arms: Combined physical exercise in water

SUMMARY:
The main objective of the study is to compare the effect of two different types of physical exercise modalities on glycated hemoglobin and blood pressure in elderly individuals with multimorbidity. The main characteristic of the proposal is that it is experimental, with two intervention groups with physical exercise that will be randomized in the order of participation of the groups and forwarded to the researchers regarding the evaluations and training periods. In addition, the study will be controlled, as it has a control group that will not perform any intervention with physical exercises during the study period. To allocate the participants in each exercise group and for the control group, the researchers will use the 1:1 method, the user will receive an automatic generator through the random.org website.

The main questions raised by the studies will be: Is land-based training more effective than aquatic training for this population in improving the primary outcomes? Is there a difference between training at these intensities and not doing any physical exercise in this population with these primary outcomes?

Participants in the 2 intervention groups will:

Train 3x per week for 10 weeks at intensities that will progress over the weeks.

ELIGIBILITY:
Inclusion Criteria:

* Being elderly adult 60 years old
* Having grade 1 medicated hypertension (systolic blood pressure ≥ 140 and diastolic blood pressure ≥ 90) or having type 2 diabetes mellitus
* Volunteers may have other morbidities such as: anxiety/depression, knee osteoarthritis or obesity
* Be fit for the practice of physical activity

Exclusion Criteria:

* Being a smoker
* Have severe musculoskeletal problems that prevent you from carrying out physical activities
* Unable to carry out the protocol completely

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin (Hb1Ac) | 10 weeks
  In the pre- and post-training moments during the morning and fasting period, venous blood samples will be collected to analyze the glycemic profile. The outcome measure will be expressed as a percentage (%), representing the average blood glucose level over the last 2 to 3 months.
Blood pressure | 10 weeks
  Office blood pressure (OBP) will be evaluated and monitored during pre-training moments using automatic monitors, and Home Blood Pressure Monitoring (HBPM) will be conducted with appropriate collection devices according to the 2021 European Society of Hypertension practice guidelines for office and out-of-office blood pressure measurement.The results of Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) will be shown in millimeters of mercury (mmHg) for OBP and HBPM.

SECONDARY OUTCOMES:
Heart rate variability | 10 weeks
  Heart rate will be monitored through a heart rate monitor (POLAR® HR monitor model RS800cx (recording frequency: 1000Hz), consequently obtaining heart rate variability, and such collection will take place in a sitting position with spontaneous breathing, for 20 minutes at total rest at the appropriated local
Lipid Profile (LDL, HDL, VLDL and Triglycerides) | 10 weeks
  In the pre- and post-training moments during the morning and fasting period, venous blood samples will be collected to analyze the lipid (LDL; HDL; VLDL; triglycerides and total cholesterol). The unit of measurement used to express the results will be mg/dL.
Body Mass Index (BMI) | 10 weeks
  The participants' body mass and height will be measured using bioimpedance and a stadiometer, respectively. Thus, researchers will have access to the BMI weight (kg)/height (m2).
Fasting glucose | 10 weeks
  In the pre- and post-training moments during the morning and fasting period, venous blood samples will be collected to analyze the glycemic profile by fasting glucose (mg/dL).
Agility | 10 weeks
  Agility and mobility will be assessed with the Timed up and go test. All testing protocol will be followed and results will be displayed as per guidelines.
Cardiorespiratory fitness | 10 weeks
  The 6-minute walk test will be performed to measure the cardiorespiratory capacity of the elderly. It will be carried out according to the proposed guidelines
Hand grip strength | 10 weeks
  The handgrip strength test will be performed with a calibrated device and the test protocol will be guided by official guidelines.
Sit and stand test | 10 weeks
  The test will measure the strength of the lower limbs of elderly people and will be guided by official guidelines
World Health Organization Quality of Life - WHOQOL questionnaire | 10 weeks
  Quality of life will be measured using the World Health Organization Quality of Life - WHOQOL questionnaire validated for the Portuguese language.The WHOQOL uses a scoring system ranging from 1 to 5, with responses varying according to the intensity, frequency, or severity of each item. The instrument is structured into four primary domains and includes several supplementary items. In the summation, the score ranges from a minimum of 4, indicating poor quality of life, to a maximum of 20, reflecting a good quality of life.
Internation Physical Activity - IPAQ questionnaire | 10 weeks
  The Internation Physical Activity - IPAQ questionnaire will measure each participant's level of physical activity. It includes items regarding the frequency, duration, and intensity of physical activity undertaken in the previous week. The summation of responses results in a total score that is categorized into low, moderate, or high levels of physical activity. Higher scores indicate greater physical activity, which correlates with enhanced physical fitness and overall health.
Pittsburgh Sleep Quality Index - PSQIquestionnaire | 10 weeks
  Sleep quality level will be measured using the Pittsburgh Sleep Quality Index -PSQI questionnaire. The questionnaire consists of 19 items that cover various dimensions of sleep, including sleep latency, duration, disturbances, efficiency, and medication use. These items are grouped into seven component scores, which are aggregated to derive a global score. The total PSQI score ranges from 0 to 21, with higher scores indicating poorer sleep quality. A global score greater than 5 typically indicates significant sleep disturbances, while lower scores reflect better sleep quality.
Depression, Anxiety, and Stress Scale - DASS 21 | 10 weeks
  Depression, anxiety and stress will be measured using a scale given by the Depression, Anxiety, and Stress Scale - DASS 21 questionnaire. The scale is composed of 21 items, divided into three subscales: depression, anxiety, and stress, each consisting of 7 items. Participants rate each item on a 4-point Likert scale, ranging from 0 (not at all) to 3 (very much or most of the time), reflecting the frequency of symptoms experienced during the previous week. Subscale scores are computed by summing the item responses within each subscale. Higher scores indicate greater severity of depression, anxiety, or stress. The resulting scores are classified into severity levels, ranging from normal to extremely severe.
Balance test | 10 weeks
  Balance will be analyzed through a biomechanical assessment with a force platform for each volunteer.
Muscle electrical activity | 10 weeks
  The electrical activity of the vastus medialis and lateralis muscles will be assessed with surface electromyography electrodes.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Gonçalves, Professor, Principal Investigator — Universidade do Porto; Victor Hugo V Carrijo, MsC. Physioterapy, Principal Investigator — Universidade do Porto; Mario Jorge O Costa, Professor, Principal Investigator — Universidade do Porto
Locations (1):
- Municipal Pavilion of Vila Nova de Famalicão, Vila Nova de Famalicão, Braga District, Portugal

IPD SHARING:
Plan to Share IPD: No